CLINICAL TRIAL: NCT02326233
Title: A Randomised, Open-labelled, Two-arm, Parallel Group, Single-dose Study to Compare the Pharmacokinetics, Safety, and Tolerability of the Pre-filled Pen and PFS of SB5 in Healthy Subjects
Brief Title: Pharmacokinetics, Safety, and Tolerability Study of the Pen and PFS of SB5 in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Samsung Bioepis Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: SB5-G12-NHV; 2014-005178-12 (EudraCT Number)
Record Dates: First submitted 2014-12-22; First posted 2014-12-29 (Estimated); Results first posted 2019-03-18 (Actual); Last update posted 2019-03-18 (Actual); Status verified 2018-12

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Pen of SB5 (Experimental): Pen of SB5, single-dose of 40 mg via subcutaneous injection (study drug)
  Interventions: Biological: Pen of SB5
- PFS of SB5 (Active Comparator): PFS of SB5, single-dose of 40 mg via subcutaneous injection (reference drug)
  Interventions: Biological: PFS of SB5

INTERVENTIONS:
Biological: Pen of SB5
  Arms: Pen of SB5
Biological: PFS of SB5
  Arms: PFS of SB5

SUMMARY:
The purpose of this study is to compare the pharmacokinetics, safety, and tolerability of the pre-filled pen and pre-filled syringe of SB5 in healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects
* Have a body mass index between 20.0 to 29.9 kg/m², inclusive.

Exclusion Criteria:

* History and/or current presence of clinical significant atopic allergy, hypersensitivity or allergic reactions, also including known or suspected clinically relevant drug hypersensitivity to any components of the test and reference investigational product formulation or comparable drugs
* Active or latent Tuberculosis or who have a history of Tuberculosis
* History of invasive systemic fungal infections or other opportunistic infections
* Systemic or local infection, a known risk for developing sepsis and/or known active inflammatory process
* Serious infection associated with hospitalisation and/or which required intravenous antibiotics
* History of and/or current cardiac disease
* Have received live vaccine(s) within 4 weeks prior to Screening or who will require live vaccine(s) between Screening and the subject's last visit
* Intake medication with a half-life > 24 h within 4 weeks or 10 half-lives of the medication prior to investigational product administration

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 190 (Actual)
Dates: Start 2015-06; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- Samsung Investigational Site, Antwerp, Belgium
- Samsung Investigational Site, Auckland, New Zealand

REFERENCES:
- [Derived] Shin D, Lee Y, Jeong D, Ellis-Pegler R. Comparative pharmacokinetics of an adalimumab biosimilar SB5 administered via autoinjector or prefilled syringe in healthy subjects. Drug Des Devel Ther. 2018 Nov 5;12:3799-3805. doi: 10.2147/DDDT.S169082. eCollection 2018. PMID 30464411

RESULTS

PARTICIPANT FLOW:
Groups:
- Pen of SB5: Pen of SB5, single-dose of 40 mg via subcutaneous injection (study drug)
  Pen of SB5
- PFS of SB5: PFS of SB5, single-dose of 40 mg via subcutaneous injection (reference drug)
  PFS of SB5
Period: Overall Study
Arm/Group | Pen of SB5 | PFS of SB5
Started | 95 | 95
Completed | 95 | 94
Not Completed | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Pen of SB5 | PFS of SB5 | Total
Number analyzed (Participants) | 95 | 95 | 190
Age, Continuous [Mean (Standard Deviation); unit: years] | 31.2 (10.58) | 30.5 (11.41) | 30.8 (10.98)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 10 | 19
  Male | 86 | 85 | 171
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 3 | 8
  Not Hispanic or Latino | 90 | 92 | 182
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 1 | 2
  Asian | 6 | 8 | 14
  Native Hawaiian or Other Pacific Islander | 1 | 4 | 5
  Black or African American | 3 | 1 | 4
  White | 78 | 80 | 158
  More than one race | 6 | 1 | 7
  Unknown or Not Reported | 0 | 0 | 0
Height (cm) [Mean (Standard Deviation); unit: cm] | 177.63 (7.753) | 177.89 (7.814) | 177.76 (7.764)

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Concentration-time Curve From Time Zero to Infinity (AUCinf)
Time Frame: 0, 24, 48, 96, 120, 144, 168, 216, 264, 336, 408, 504, 600, 696, 840, 1008, and 1344 h postdose
Measure: Mean (Standard Deviation); unit: h·μg/mL
Arm/Group | Pen of SB5 | PFS of SB5
Number analyzed (Participants) | 94 | 94
h·μg/mL | 2743.2 (1081.76) | 2503.3 (1043.69)

2. Primary Outcome: Area Under the Concentration-time Curve From Time Zero to the Last Quantifiable Concentration (AUClast)
Time Frame: 0, 24, 48, 96, 120, 144, 168, 216, 264, 336, 408, 504, 600, 696, 840, 1008, and 1344 h postdose
Measure: Mean (Standard Deviation); unit: h·μg/mL
Arm/Group | Pen of SB5 | PFS of SB5
Number analyzed (Participants) | 94 | 94
h·μg/mL | 2329.2 (733.30) | 2182.2 (724.98)

3. Primary Outcome: Maximum Serum Concentration (Cmax)
Time Frame: 0, 24, 48, 96, 120, 144, 168, 216, 264, 336, 408, 504, 600, 696, 840, 1008, and 1344 h postdose
Measure: Mean (Standard Deviation); unit: μg/mL
Arm/Group | Pen of SB5 | PFS of SB5
Number analyzed (Participants) | 94 | 94
μg/mL | 3.803 (1.0697) | 3.673 (0.8810)

4. Secondary Outcome: Time to Reach Cmax (Tmax)
Time Frame: 0, 24, 48, 96, 120, 144, 168, 216, 264, 336, 408, 504, 600, 696, 840, 1008, and 1344 h postdose
Measure: Median (Full Range); unit: h
Arm/Group | Pen of SB5 | PFS of SB5
Number analyzed (Participants) | 94 | 94
h | 168.000 [24.00 to 504.12] | 168.000 [48.00 to 408.00]

ADVERSE EVENTS:
Arm/Group | Pen of SB5 | PFS of SB5
Serious Adverse Events (participants affected / at risk) | 1/95 | 2/94
Other Adverse Events (participants affected / at risk) | 39/95 | 28/94
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pen of SB5 (N=95) | PFS of SB5 (N=94)
Clavicle fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Hand fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Schizophrenia (Psychiatric disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pen of SB5 (N=95) | PFS of SB5 (N=94)
Fatigue (General disorders) | 7 (7) | 1 (1)
Vessel puncture site bruise (General disorders) | 5 (5) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 15 (15) | 18 (19)
Back pain (Musculoskeletal and connective tissue disorders) | 6 (7) | 1 (1)
Headache (Nervous system disorders) | 6 (6) | 8 (10)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes